CLINICAL TRIAL: NCT07023354
Title: Open Label, Single Dose, Parallel-group Study to Evaluate the PK and the Safety and Tolerability of Single Oral Doses of BI 1291583 in Trial Participants With Mild, Moderate and Severe Hepatic Impairment as Compared to Matched, Hepatically Healthy Trial Participants.
Brief Title: A Study to Test How BI 1291583 is Taken up in the Blood of People With and Without Liver Problems
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1397-0024; U1111-1312-8762 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-06-10; First posted 2025-06-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Hepatic Impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: Participants with mild liver impairment (Experimental): Child-Pugh classification A; score of 5 - 6 points.
  The Child-Pugh score assesses chronic liver disease severity, factoring in three lab parameters (total bilirubin, serum albumin, and prothrombin time), ascites, and hepatic encephalopathy. Scores are categorized as follows: 5-6 (Class A, mild), 7-9 (Class B, moderate), and 10-15 (Class C, severe), with higher scores indicating more severe disease.
  Interventions: Drug: BI 1291583
- Group 2: Participants with moderate liver impairment (Experimental): Child-Pugh classification B; score of 7 - 9 points.
  The Child-Pugh score assesses chronic liver disease severity, factoring in three lab parameters (total bilirubin, serum albumin, and prothrombin time), ascites, and hepatic encephalopathy. Scores are categorized as follows: 5-6 (Class A, mild), 7-9 (Class B, moderate), and 10-15 (Class C, severe), with higher scores indicating more severe disease.
  Interventions: Drug: BI 1291583
- Group 3: Participants with severe liver impairment (Experimental): Child-Pugh classification C; score of 10-15 points.
  The Child-Pugh score assesses chronic liver disease severity, factoring in three lab parameters (total bilirubin, serum albumin, and prothrombin time), ascites, and hepatic encephalopathy. Scores are categorized as follows: 5-6 (Class A, mild), 7-9 (Class B, moderate), and 10-15 (Class C, severe), with higher scores indicating more severe disease.
  Interventions: Drug: BI 1291583
- Group 4: Healthy trial participants with normal liver function (Experimental): Matched to 8 demographic clusters generated from the 24 trial participants of Groups 1 through 3.
  Interventions: Drug: BI 1291583

INTERVENTIONS:
Drug: BI 1291583 — BI 1291583
  Other Names: Verducatib

SUMMARY:
This study is open to adults aged between 18 and 80 years of age with a body mass index (BMI) of 18.5 to 42 kg/m². People with or without liver problems can take part in the study. The purpose of this study is to find out how much of a medicine called BI 1291583 gets into the blood of people with and without liver problems. BI 1291583 is being developed to treat people with bronchiectasis, a chronic disease of the lungs. People living with this condition often also have liver problems. Therefore, it is important to find out whether liver problems influence the amount of BI 1291583 that gets into the blood.

Study participants receive a single dose of BI 1291583 as a tablet taken by mouth. Participants are divided into 4 groups based on how well their liver works: 1 group without liver problems, and 3 groups with mild, moderate, and severe liver problems. Each participant without liver problems is matched with participants from the other groups based on factors such as age, sex, smoking habits, and body weight to ensure accurate comparisons.

Participants are in the study for about 3 months. They stay for 3 days at the study site and also visit the study site up to 9 times. During these visits, the doctors collect information about participants' health. To assess the study endpoints, the doctors regularly take blood samples from the participants. The doctors regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria :

1. Male or female trial participants aged ≥18 and ≤80 years at screening
2. Body Mass Index (BMI) of 18.5 to 42 kg/m² (inclusive)
3. Signed and dated written informed consent in accordance with International Council on Harmonisation (ICH) Harmonized Guideline for Good Clinical Practice (GCP) and local legislation prior to admission to the trial
4. Female trial participants who meet any of the following criteria for a highly effective contraception from at least 30 days before the first administration of trial medication until 5 months after trial dosing

   * Use of combined (oestrogen and progestogen containing) hormonal contraception that prevents ovulation (oral, intravaginal or transdermal), plus condom
   * Use of progestogen-only hormonal contraception that inhibits ovulation (only injectables or implants), plus condom
   * Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS) plus use of condom
   * Sexually abstinent
   * A vasectomised sexual partner who received medical assessment of the surgical success (documented absence of sperm) and provided that partner is the sole sexual partner of the trial participant
   * Surgically sterilised (including hysterectomy) plus use of condom
   * Postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with levels of Follicle Stimulating Hormone (FSH) above 25 U/L and oestradiol below 30 ng/L is confirmatory)

In addition to the overall inclusion criteria given, trial participants with impaired hepatic function must fulfil the following criteria:

1. Hepatic impairment classified as Child-Pugh A (score 5-6 points) or Child-Pugh B (score 7-9 points) or Child Pugh C (score 10-15 points)
2. Absence of significant abnormalities, as based on a complete medical history including a full physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests at both screening and admission to trial site, with the exception of findings that in the opinion of the investigator are consistent with the participant's hepatic impairment
3. Medication and/or treatment regimens must have been stable (i. e., no dose adjustments) for at least 7 days or 5 half-lives (whichever is longer) prior to the planned randomisation and should be kept stable until study completion. Fluctuating treatment regimens may be considered for inclusion on a case-by-case basis if the underlying disease is under control in the opinion of the investigator and must be agreed to by both the investigator and the sponsor's medical monitor

In addition to the overall inclusion criteria given, trial participants with normal hepatic function must fulfill the following criteria:

1. Individually matched to trial participation with hepatic impairment according to sex, age, smoking habit and weight

Exclusion Criteria:

Exclusion criteria applying to all trial participants:

1. Any medical condition or finding in the medical examination that in the investigator's opinion assessed as clinically relevant, poses a safety risk for the trial participant or may interfere with the study objectives (except for conditions associated with hepatic impairment in trial participant with compromised hepatic function)
2. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance (apart from values due to underlying disease)
3. Severe gastrointestinal, renal (estimated Glomerular Filtration Rate (eGFR) Chronic Kidney Disease Epidemiology (CKD-EPI) <40 ml/min/1.73 m2 for the hepatic impaired trial participants and Estimated Glomerular Filtration Rate (eGFR) Chronic Kidney Disease Epidemiology (CKD-EPI) <60 ml/min/1.73 m2 for matched controls), respiratory, cardiovascular, metabolic, immunological or hormonal disorders assessed as clinically relevant by the Investigator
4. Alpha fetoprotein >50 ng/mL (>50 µg/L) at screening
5. Surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except cholecystectomy, appendectomy or simple hernia repair)
6. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
7. History of relevant orthostatic hypotension, fainting spells, or blackouts
8. Relevant chronic or acute infections
9. Further exclusion criteria apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2026-07-04 (Estimated); Study Completion 2026-07-04 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 672 h (AUC0-672h) | Up to Day 29
Maximum measured concentration of the analyte in plasma (Cmax) | Up to Day 29

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞ of BI 1291583) | Up to Day 29
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz of BI 1291583) | Up to Day 29

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Orlando Clinical Research Center, Orlando, Florida
  - Tranquil Clinical Research, Houston, Texas
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com